CLINICAL TRIAL: NCT05223556
Title: Investigation of the Accuracy of a Self-testing Diagnosis Imaging Model for Diabetic Retinopathy
Brief Title: Self-testing Diagnosis Imaging Model for Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020KYPJ201
Record Dates: First submitted 2022-01-22; First posted 2022-02-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shaoguan Diabetic cohort: Patients with diabetes ages 30-80 were enrolled in Shaoguan Diabetic Eye Screening Programme, who will receive diabetic retinopathy screening both in a remote diagnostic imaging site and in a tertiary hospital
  Interventions: Device: Full Self-Diagnostic device in a remote diagnostic imaging site; Device: Human imager operated diagnostic device in the hospital

INTERVENTIONS:
Device: Full Self-Diagnostic device in a remote diagnostic imaging site — Full Self-Diagnostic CRP+OCT imaging, followed by online consultation
Device: Human imager operated diagnostic device in the hospital — Human imager operated CRP imaging with dilated pupils, followed by face-to-face consultation

SUMMARY:
This is a prospective clinical study. At the Shaoguan Diabetic Eye Screening Programme, patients ages 30-80 will undergo the two diagnostic models: (1) in a remote diagnostic clinic site, patients undergo a self-testing device that provides both color retinal photography (CRP) and optical coherence tomography (OCT) imaging of nondilated pupils, and receive an online consultation provided by a retinal specialist; (2) on a separate day, patients visit the tertiary hospital, undergo traditional imaging of dilated pupils acquired by a non-expert imager using a traditional CRP imaging device at the point of care, and receive a face-to-face consultation provided by a retinal specialist.

Within one week of receiving both diagnostic imaging services, patient preferences are assessed and they decide which diagnostic imaging model is preferred.

ELIGIBILITY:
Inclusion Criteria:

1. who are enrolled in the Shaoguan Diabetic Eye Screening Programme for their eye check-up
2. who are diagnosed with diabetes and aged between 30 years and 80 years
3. be able to sit for an imaging device for image acquisition
4. be capable of giving their own consent

Exclusion Criteria:

1. who are pregnant or nursing women

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants from Shaoguan diabetic cohort
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Accuracy in the diagnosis of referral retinal lesions | 1 week
  Accuracy in the diagnosis of referral retinal lesions using the self-testing diagnosis imaging

SECONDARY OUTCOMES:
The agreement between the two modalities | 1 week
  kappa value to assess the agreement between the two modalities in the diagnosis of referral retinal lesions
Feasibility of self-testing diagnosis imaging model | 1 week
  Feasibility is measured by examination completion rate
Feasibility of self-testing diagnosis imaging model | 1 week
  Feasibility is measured by interpretable image rate
Satisfaction of participants as measured by questionnaire | 1 week
  Satisfaction is measured by a questionnaire between the two modalities

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No